CLINICAL TRIAL: NCT02102191
Title: Acute Physiological Effects of Electronic Sigarette vs Cigarette Smoking: a RCT
Brief Title: Acute Physiological Effects of Electronic Sigarette vs Cigarette Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: Fondazione Salvatore Maugeri (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, professor of respiratory disease, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 972CE; 23 (Other: SIME)
Record Dates: First submitted 2014-03-27; First posted 2014-04-02 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Individuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cigarette (Active Comparator): common cigarette sold in the stores
  Interventions: Device: e-cigarette; Device: cigarette
- e-cigarette (Active Comparator): e-cigarette (Ovale Elips)
  Interventions: Device: e-cigarette; Device: cigarette

INTERVENTIONS:
Device: e-cigarette — smoking cigarette without tobacco
Device: cigarette — smoking cigarette with tobacco

SUMMARY:
Because e-cigarettes do not contain or burn tobacco, they do not appear to deliver the known toxins found in conventional cigarette smoke.However e-Cigarettes with low dose of tobacco were found to have immediate adverse physiologic effects after short-term use that are similar to some of the effects seen with tobacco smoking.

In this study we wanted to assess the short-time effect of one e-cigarette with no tobacco vs a "traditional" cigarette.

10 n-smoking subject and 10 actual smokers will be enrolled in the randomized trial.

DETAILED DESCRIPTION:
On day 1 the subjects will be asked to smoke either the e-cigarette or a "traditional" one for 5 minutes. On day 2 the subject will be ask to smoke for 5 minutes the other kind of cigarette.

Exhaled Nitric Oxide will be measured in a sitting position with a nose clip using an analyzer equipped with a software program. The patient will be instructed to inhale as deeply as possible to total lung capacity through a filter mouthpiece and consecutively exhale at a mouth fl ow rate of 50 mL/s for 10 s. Three consecutive trials will be performed with a 30-s interval.

Dynamic Lung Volumes: Flows and lung volumes will be measured in the sitting position, a spirometry system (heated pneumotach, with the highest FEV 1 recorded in line with pulmonary guidelines. Spirometry will be measured according to the recommendations of the American Thoracic Society/European Respiratory Society task force guidelines. FEV 1, FVC, FEV 1 %, peak expiratory fl ow (PEF), and maximal expiratory fl ow (MEF) at 25%, 50%, and 75% of vital capacity will be measured. Each maneuver will be repeated for at least three technically acceptable forced expiratory fl ow curves.

ELIGIBILITY:
Inclusion Criteria:

* 10 no smoking healthy individuals
* 10 smoking (>20 pack/yr) healthy individuals

Exclusion Criteria:

* pre-existing diseases
* FEV1/FVC ratio<70%

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
spirometric data | five minutes

SECONDARY OUTCOMES:
nitric oxyde level | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: stefano nava, md, Study Chair — AO Sant'Orsola
Locations (1):
- Fondazione Salvatore Maugeri, Pavia, Province, Italy

REFERENCES:
- [Derived] Ferrari M, Zanasi A, Nardi E, Morselli Labate AM, Ceriana P, Balestrino A, Pisani L, Corcione N, Nava S. Short-term effects of a nicotine-free e-cigarette compared to a traditional cigarette in smokers and non-smokers. BMC Pulm Med. 2015 Oct 12;15:120. doi: 10.1186/s12890-015-0106-z. PMID 26459355